CLINICAL TRIAL: NCT05927701
Title: Self-perceived Health Status and Healthcare Consumption of Idiopathic Scoliosis Patients Treated More Than 20 Years Ago: How Much do Operated and Non-operated Patients Differ?
Acronym: HISTORY
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8867
Record Dates: First submitted 2023-06-22; First posted 2023-07-03 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Adolescent Idiopathic Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-Surgical Group: Patients treated non-surgically during adolescence (<18 years of age) with a baseline Cobb >40º and minimum 20 years of follow-up.
  Interventions: Other: Group comparaison
- Surgical Group: Patients treated surgically during adolescence (<18 years of age) with a baseline Cobb >40º, and minimum 20 years of follow-up
  Interventions: Other: Group comparaison

INTERVENTIONS:
Other: Group comparaison — Questionnaires

SUMMARY:
Adolescent idiopathic scoliosis (AIS) is a common condition that affects millions of patients worldwide. This is characterized by a spinal deformity that leads to a deformation of the trunk, an imbalance of the shoulders and waist folds as well as the appearance of gibbosity.

Posterior arthrodesis correction is a common practice surgery for the treatment of AIS after failure of medical treatment with a corset or functional rehabilitation. Surgery allows functional improvement and is indicated for curves greater than medically treated scoliosis.

The objective of this international study is to have a better understanding of the long-term outcomes (> 20 years of follow-up) after treatment (surgical and non-surgical) of AIS and to compare the long-term status of the patient with AIS to the general population of the same age, sex and comorbidities.

All of this information will help justify or modify the strategy, techniques and goals of early treatment in adolescence to achieve a better long-term outcome.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Adolescent Idiopathic Scoliosis
* Main baseline curve magnitude over 40º
* Aged 10 to 18 years at the time of treatment (surgical or nonsurgical)
* More than 20 years of follow up
* Current contact information available

Exclusion Criteria:

* Non-idiopathic scoliosis
* Younger than 10 or older than 18 at the time of initial treatment
* Less than 20 years of follow up
* Patients unable to understand and answer the questionnaires because of language difficulties or because of cognitive impairments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a Diagnosis of Adolescent Idiopathic Scoliosis aged 10 to 18 years at the time of treatment (surgical or nonsurgical)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2026-07-06 (Estimated); Study Completion 2026-07-06 (Estimated)

PRIMARY OUTCOMES:
Long-term quality of life | 1 day
  Evaluate from the specific questionnaire for vertebral deformities: Scoliosis Research Society revisited(SRS-22r) (scale 0-5) with 5 sub-domains,higher scores representing greater patient quality of life.

SECONDARY OUTCOMES:
The long-term quality of life | 1 day
  Assess the long-term quality of life (> 20 years), health status, and social and demographic outcomes of adult patients who underwent treatment (surgical and non-surgical) for idiopathic scoliosis during adolescence by the questionnaire EQ-5D-5L (100 is the best health you can imagine.
  0 is the worst health you can imagine)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Clinique du dos, Bruges
  - Hôpitaux Universitaires de Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: Undecided